CLINICAL TRIAL: NCT00286026
Title: Azithromycin in Control of Trachoma II
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Prevalence of infection for screened population too low (<7%) to enroll anyone.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Julius Schachter, Professor of Laboratory Medicine, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H1079-17254; 5R01AI048789 (NIH)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Trachoma
Keywords: Chlamydia trachomatis
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Subjects residing in villages assigned to treatment arm 1 will receive a clinical evaluation for trachoma and provide a swab specimen of conjunctivae of the R eye at enrollment (Day 0); will be treated with Azithromycin at Day 30; will be re-screened (clinical evaluation and swab specimen of R eye collected) at Day 60; and again at Day 360.
  Interventions: Drug: Azithromycin
- Arm 2 (Experimental): Subjects residing in villages assigned to treatment arm 2 will receive a clinical evaluation for trachoma and provide a swab specimen of conjunctivae of the R eye at enrollment (Day 0), as well as receive an initial treatment with Azithromycin; will receive a second dose of Azithromycin at Day 30; will be re-screened (clinical evaluation and swab specimen of R eye collected) at Day 60; and again at Day 360.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 1 gm Azithromycin orally, provided as four 250 mg tablets for adults; pediatric suspension will be provided to children > 1 year old (20 mg/kg body weight) to a maximal dose of 500 mg. One dose vs 2 doses given 30 days apart.
  Other Names: Zithromax; Zmax

SUMMARY:
Trachoma is the world's leading cause of preventable blindness. This disease, caused by Chlamydia trachomatis, is endemic in many parts of the developing world. In 1990s we evaluated the use of community-wide treatment with oral azithromycin in a project called Azithromycin in Control of Trachoma (ACT). This approach resulted in clinical improvement and dramatic reduction in prevalence of chlamydial infection through a 1-year follow-up. We enrolled the ACT villages, as well as an additional village that had not had any prior treatments, in our ACT II (2005) study and performed clinical surveys to assess trachoma activity testing conjunctival swabs for the presence of C. trachomatis by nucleic acid amplification tests (NAATs). Thus, we hoped to determine the long-term (10 year) effects of azithromycin treatment.

We have completed the census and clinical survey of the initial three villages. Mass treatment with azithromycin would not be justified with such low rates (1.8 - 4%) of ocular chlamydial infection. We have treated only those living in households with one or more cases of chlamydial infection and we will not follow up on these individually treated families.

In order to achieve the goals of our study, we now propose to identify other more remote villages with trachoma infection rates of 20% or more to evaluate the effect of community-wide treatment with single dose of oral azithromycin. If one or more of these villages (dependent upon population) has trachoma rates of 20% or more they will be invited to participate in the azithromycin treatment. In one set of subjects (1 or 2 villages, dependent upon population and infection rate) we will perform treatment, and follow them up at 2-, 12-, and 24-months post-treatment to ascertain infection rates. In a second set of subjects (1 or 2 villages, dependent upon population and infection rate) we will perform treatment, then perform re-treatment at 30-days post initial treatment, and follow them up at 2-, 12-, and 24-months post-treatment to ascertain infection rates. This should help us determine the need for/and the best time for re-treatment to eliminate blinding trachoma, as some recent studies suggest there is a 2-4% failure rate in the initial treatment. In sum, this study should provide a rational approach to use of community-wide azithromycin treatment to eliminate blinding trachoma as a public health problem

DETAILED DESCRIPTION:
This is operational research aimed at better defining the use of oral azithromycin as part of the SAFE strategy to eliminate blinding trachoma.

1. Before the examinations, we will do a census and a sketch map of houses in each village. Particular emphasis will be placed on identifying all the children between 1 and 6 years of age. These children are the chief reservoir of infection, and would have been too young (or unborn) at the ACT study treatment, so it is of particular interest to determine their disease and infection status.
2. Egyptian ophthalmologists will examine the eyelids, conjunctiva and cornea using magnifying loupes and a hand held light, with grading following the ACT protocol which contains categories referable to the W.H.O. detailed grading scheme. The clinical findings will be recorded on a standardized form.
3. Egyptian health aides will photograph the inside of the right upper eyelid of all subjects. The photographs of the subjects at the initial visit and all subsequent examinations will be examined to confirm the consistency of clinical findings over the period of the study.
4. To test for chlamydial infection, a single fiber-tipped swab will be stroked gently over the conjunctiva of the right eye by an Egyptian ophthalmologist. These swabs will be placed in special tubes and tested for Chlamydia trachomatis by a nucleic acid amplification assay. [APTIMA® Gen-Probe Inc. (San Diego, CA.)] The APTIMA® assay detects DNA via r-RNA by a process called transcription mediated amplification. Laboratory testing will be performed at the Chlamydia Research Laboratory at University of California, San Francisco.
5. After the results are obtained from the nucleic acid amplification testing performed at the laboratory in San Francisco, treatment for trachoma will be done with a single-dose of oral azithromycin (20 mg/kg body weight in children, 1.0 gm adults). The azithromycin will be donated by Pfizer International. Young children will be weighed to determine the dose of azithromycin and the doses administered by a health aide under direct supervision of an Egyptian physician (Dr. Mahfouz). One set of subjects (1 or 2 villages depending upon population size, in order to generate meaningful numbers) will receive an initial treatment of 1.0 gm azithromycin; while the second set of subjects will receive an initial treatment of 1.0 gm azithromycin, followed by a second dose of 1.0 gm azithromycin at 30 days post treatment.

   1. If the prevalence of clinical trachoma is over 20% in children 10 and under, everyone in the village will be treated with oral azithromycin.

      After initial azithromycin treatment, follow-up examinations and specimen collection will be done 2, 12, and 24 months post-treatment for trachoma and chlamydial infection.
   2. If the prevalence is 10% to 20%, all children 10 and under, and the families of those children with active trachoma, will be treated.

      After initial azithromycin treatment, follow-up examinations and specimen collection will be done 2, 12, and 24 months post-treatment for trachoma and chlamydial infection.
   3. If the prevalence is less than 10%, only children with active disease and their families will receive treatment. There will be no follow-up examinations.

   Adults and older children will be told that azithromycin can cause nausea, vomiting, or loose stools or vomiting in some children and adults, and can occur in up to 5% (1 person in 20) of those treated.

   It should be noted that in our previous ACT study, more than 8,000 people received azithromycin with no complaints beyond minor gastro-intestinal upset.
6. All positive specimens will have the major outer membrane gene amplified and sequenced. The genovars will be mapped for location within villages and families and then their distribution will be followed over time, after treatment to provide a better understanding of the epidemiology of the infection. Results of the study will be used as data input for the generation of mathematical models to predict whether community-wide retreatment (or alternate strategies) will be needed, and the optimal timing for such retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Person resides within a selected rural village in a trachoma-endemic area of Egypt.

Exclusion Criteria:

* Person does not reside in one of the three rural villages being studied.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2007-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Infection with Chlamydia trachomatis diagnosed by use of NAAT | One-year

CONTACTS AND LOCATIONS:
Overall Officials: Julius Schachter, PhD, Principal Investigator — University of California, San Francisco; Chandler R Dawson, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Mabey D, Fraser-Hurt N. Antibiotics for trachoma. Cochrane Database Syst Rev. 2002;(1):CD001860. doi: 10.1002/14651858.CD001860. PMID 11869610
- [Background] Burton MJ, Frick KD, Bailey RL, Bowman RJ. Azithromycin for the treatment and control of trachoma. Expert Opin Pharmacother. 2002 Feb;3(2):113-20. doi: 10.1517/14656566.3.2.113. PMID 11829725
- [Background] Dawson CR, Schachter J. Should trachoma be treated with antibiotics? Lancet. 2002 Jan 19;359(9302):184-5. doi: 10.1016/S0140-6736(02)07463-9. No abstract available. PMID 11812548
- [Background] Bain DL, Lietman T, Rasmussen S, Kalman S, Fan J, Lammel C, Zhang JZ, Dawson CR, Schachter J, Stephens RS. Chlamydial genovar distribution after community wide antibiotic treatment. J Infect Dis. 2001 Dec 15;184(12):1581-8. doi: 10.1086/324661. Epub 2001 Dec 3. PMID 11740734
- [Background] Pechere JC. New perspectives on macrolide antibiotics. Int J Antimicrob Agents. 2001;18 Suppl 1:S93-7. doi: 10.1016/s0924-8579(01)00393-4. PMID 11574203
- [Background] Fraser-Hurt N, Bailey RL, Cousens S, Mabey D, Faal H, Mabey DC. Efficacy of oral azithromycin versus topical tetracycline in mass treatment of endemic trachoma. Bull World Health Organ. 2001;79(7):632-40. PMID 11477966
- [Background] Tabbara KF. Trachoma: a review. J Chemother. 2001 Apr;13 Suppl 1:18-22. doi: 10.1080/1120009x.2001.11782323. PMID 11434524
- [Background] Treadway G. Azithromycin: a new 15-membered macrolide. Jpn J Antibiot. 2001 Feb;54 Suppl A:70-6. PMID 11296412
- [Background] Bailey R, Lietman T. The SAFE strategy for the elimination of trachoma by 2020: will it work? Bull World Health Organ. 2001;79(3):233-6. Epub 2003 Jul 7. PMID 11285668
- [Background] Frick KD, Lietman TM, Holm SO, Jha HC, Chaudhary JS, Bhatta RC. Cost-effectiveness of trachoma control measures: comparing targeted household treatment and mass treatment of children. Bull World Health Organ. 2001;79(3):201-7. Epub 2003 Jul 7. PMID 11285663
- [Background] Holm SO, Jha HC, Bhatta RC, Chaudhary JS, Thapa BB, Davis D, Pokhrel RP, Yinghui M, Zegans M, Schachter J, Frick KD, Tapert L, Lietman TM. Comparison of two azithromycin distribution strategies for controlling trachoma in Nepal. Bull World Health Organ. 2001;79(3):194-200. Epub 2003 Jul 7. PMID 11285662
- [Background] Lietman T, Fry A. Can we eliminate trachoma? Br J Ophthalmol. 2001 Apr;85(4):385-7. doi: 10.1136/bjo.85.4.385. No abstract available. PMID 11264123
- [Background] Duran JM, Amsden GW. Azithromycin: indications for the future? Expert Opin Pharmacother. 2000 Mar;1(3):489-505. doi: 10.1517/14656566.1.3.489. PMID 11249533
- [Background] Solomon AW, Akudibillah J, Abugri P, Hagan M, Foster A, Bailey RL, Mabey DC. Pilot study of the use of community volunteers to distribute azithromycin for trachoma control in Ghana. Bull World Health Organ. 2001;79(1):8-14. Epub 2003 Nov 5. PMID 11217675
- [Background] West S. The red eye. N Engl J Med. 2000 Nov 23;343(21):1577. doi: 10.1056/NEJM200011233432117. No abstract available. PMID 11184764
- [Background] Bowman RJ, Sillah A, Van Dehn C, Goode VM, Muqit MM, Johnson GJ, Milligan P, Rowley J, Faal H, Bailey RL. Operational comparison of single-dose azithromycin and topical tetracycline for trachoma. Invest Ophthalmol Vis Sci. 2000 Dec;41(13):4074-9. PMID 11095598
- [Background] Guzey M, Aslan G, Ozardali I, Basar E, Satici A, Karadede S. Three-day course of oral azithromycin vs topical oxytetracycline/polymyxin in treatment of active endemic trachoma. Jpn J Ophthalmol. 2000 Jul-Aug;44(4):387-91. doi: 10.1016/s0021-5155(00)00167-2. PMID 10974295
- [Background] Laming AC, Currie BJ, DiFrancesco M, Taylor HR, Mathews JD. A targeted, single-dose azithromycin strategy for trachoma. Med J Aust. 2000 Feb 21;172(4):163-6. doi: 10.5694/j.1326-5377.2000.tb125541.x. PMID 10772587
- [Background] Chern KC, Shrestha SK, Cevallos V, Dhami HL, Tiwari P, Chern L, Whitcher JP, Lietman TM. Alterations in the conjunctival bacterial flora following a single dose of azithromycin in a trachoma endemic area. Br J Ophthalmol. 1999 Dec;83(12):1332-5. doi: 10.1136/bjo.83.12.1332. PMID 10574809
- [Background] Whitty CJ, Glasgow KW, Sadiq ST, Mabey DC, Bailey R. Impact of community-based mass treatment for trachoma with oral azithromycin on general morbidity in Gambian children. Pediatr Infect Dis J. 1999 Nov;18(11):955-8. doi: 10.1097/00006454-199911000-00003. PMID 10571428
- [Background] Mabey D, Bailey R. Eradication of trachoma worldwide. Br J Ophthalmol. 1999 Nov;83(11):1261-3. doi: 10.1136/bjo.83.11.1261. No abstract available. PMID 10535853
- [Background] Dawson CR. Acceptance of Medaille d'Or du Trachome by Dr. Chandler R. Dawson M. D. Kyoto, 16 May 1978. Rev Int Trach Pathol Ocul Trop Subtrop. 1978;55(3-4):21-2, 30-1. No abstract available. English, French. PMID 33432
- [Background] Schachter J, West SK, Mabey D, Dawson CR, Bobo L, Bailey R, Vitale S, Quinn TC, Sheta A, Sallam S, Mkocha H, Mabey D, Faal H. Azithromycin in control of trachoma. Lancet. 1999 Aug 21;354(9179):630-5. doi: 10.1016/S0140-6736(98)12387-5. PMID 10466664
- [Background] Chidambaram JD, Alemayehu W, Melese M, Lakew T, Yi E, House J, Cevallos V, Zhou Z, Maxey K, Lee DC, Shapiro BL, Srinivasan M, Porco T, Whitcher JP, Gaynor BD, Lietman TM. Effect of a single mass antibiotic distribution on the prevalence of infectious trachoma. JAMA. 2006 Mar 8;295(10):1142-6. doi: 10.1001/jama.295.10.1142. PMID 16522834
- [Background] West SK, Munoz B, Mkocha H, Holland MJ, Aguirre A, Solomon AW, Foster A, Bailey RL, Mabey DC. Infection with Chlamydia trachomatis after mass treatment of a trachoma hyperendemic community in Tanzania: a longitudinal study. Lancet. 2005 Oct 8;366(9493):1296-300. doi: 10.1016/S0140-6736(05)67529-0. PMID 16214600
- [Background] Mabey D, Fraser-Hurt N, Powell C. Antibiotics for trachoma. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001860. doi: 10.1002/14651858.CD001860.pub2. PMID 15846624
- [Background] Solomon AW, Holland MJ, Alexander ND, Massae PA, Aguirre A, Natividad-Sancho A, Molina S, Safari S, Shao JF, Courtright P, Peeling RW, West SK, Bailey RL, Foster A, Mabey DC. Mass treatment with single-dose azithromycin for trachoma. N Engl J Med. 2004 Nov 4;351(19):1962-71. doi: 10.1056/NEJMoa040979. PMID 15525721